CLINICAL TRIAL: NCT06002360
Title: The Effect of Reach Out and Read on Home Literacy Scores, Parental Stress, and Parent-Infant Bonding in the Neonatal ICU
Brief Title: Reach Out and Read (ROR) in the Neonatal Intensive Care Unit (NICU) Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Devin McKissic, Fellow, Neonatology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00015592
Record Dates: First submitted 2023-08-15; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Anxiety; Parent-Child Relations; Literacy
MeSH Terms: conditions — Anxiety Disorders; Literacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reach Out and Read (Experimental): Families assigned to this group will receive Reach Out and Read education every two weeks between enrollment and when their infant reaches 36 weeks gestation.
  Interventions: Behavioral: Reach Out and Read
- Control (No Intervention): Standard neonatal care

INTERVENTIONS:
Behavioral: Reach Out and Read — Families will be provided with a book and ROR programming from trained study team members (either the principal investigator or a research assistant, both of whom are ROR trained). ROR programming will include discussion of current reading practices, anticipatory guidance on the importance and benefits of reading, modeling of active reading, discussion of how to incorporate reading into a daily routine and answering any questions parents/caregivers may have.
  Arms: Reach Out and Read

SUMMARY:
The goal of this clinical trial is to learn about the effects of the Reach Out and Read program on infants and their families in the neonatal ICU. The main goals of this study are:

* To complete a needs assessment for literacy interventions in the NICU population through evaluating baseline home literacy scores.
* To evaluate the effects of the ROR intervention on parental stress levels as assessed by the 6-question State-Trait Anxiety Index (STAI-6)
* To evaluate the effects of the ROR intervention on parent-infant bonding by comparing scores on the 25-item Postpartum Bonding Questionnaire (PBQ)
* To evaluate the effects of the ROR intervention on the home literacy environment by comparing home literacy scores

Participants will complete three questionnaires that include demographic information, home literacy scores, the Postpartum Bonding Questionnaire and the State-Trait Anxiety Index; once at study enrollment, once at 36 weeks corrected gestational age, and once at 3 months corrected gestational age.

Researchers will compare the control group (standard care) and a group that receives Reach Out and Read education to see whether exposure to Reach Out and Read affects literacy behaviors, parental anxiety, and parent-infant bonding.

ELIGIBILITY:
Inclusion Criteria:

* Families of subjects born between 24w0d and 33w6d gestation
* Primary language is English or Spanish

Exclusion Criteria:

* Severe clinical instability such that the principal investigators do not think the infant will survive to 36 weeks gestation

Max Age: 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effects of the ROR intervention on the home literacy environment by comparing home literacy scores | Between enrollment and 3 months corrected gestational age for infant
To evaluate the effects of the ROR intervention on parental stress levels as assessed by the 6-question State-Trait Anxiety Index (STAI-6) | Between enrollment and 3 months corrected gestational age for infant
To evaluate the effects of the ROR intervention on parent-infant bonding by comparing scores on the 25-item Postpartum Bonding Questionnaire (PBQ) | Between enrollment and 3 months corrected gestational age for infant
To complete a needs assessment for literacy interventions in the NICU population through evaluating baseline home literacy scores. | At enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Devin McKissic, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center NICU, Seattle, Washington, United States